CLINICAL TRIAL: NCT06073106
Title: Targeting Osteosarcopaenia and Multimorbidity for Frailty Prevention Through Identification and Deep Phenotyping Methods in Healthy Aging and High-burden Disease Cohorts.
Brief Title: Targeting Osteosarcopaenia and Multimorbidity for Frailty Prevention
Acronym: OPTIMA-C
Status: Recruiting | Type: Observational
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: Rehabilitation Research Institute of Singapore (RRIS) (Unknown); Woodlands Health (WH) (Unknown)
Responsible Party: Sponsor
Other Study IDs: DSRB 2023/00105
Record Dates: First submitted 2023-09-20; First posted 2023-10-10 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Stroke; Traumatic Brain Injury; Knee Osteoarthritis; Breast Cancer
Keywords: Frailty; Multimorbidity; Osteosarcopaenia
MeSH Terms: conditions — Stroke; Brain Injuries, Traumatic; Osteoarthritis, Knee; Breast Neoplasms; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood samples will be collected (50ml; about 10 teaspoons) for lab assay to assess metabolic health and inflammation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Stroke: Both acutely admitted stroke patients undergoing rehabilitation and chronic recovered stroke outpatients will be recruited.
- Traumatic Brain Injury: Both acutely admitted TBI patients undergoing rehabilitation and chronic recovered TBI outpatients will be recruited.
- Breast Cancer: Only recovered breast cancer patients.
- Knee Osteoarthritis: For patients with chronic knee osteoarthritis.

SUMMARY:
The aging population and its accompanying burden from non-communicable chronic diseases predicts an increasing impact imposed by frailty on healthcare systems. This is due to a lack of normative data for older adults and reliable risk stratification methods to develop effective approaches to the prevention of frailty.

In this study, the investigators plan to form a common dataset for phenotype identification, risk stratification of frailty and its targeted treatment plans in the at-risk and mildly frail population.

DETAILED DESCRIPTION:
Osteosarcopaenia and multimorbidity have emerged as two key antecedent factors driving the cycle of frailty, leading to adverse outcomes. However, it remains unclear how multimorbidity and/or osteosarcopaenia act singly or in concert to influence the expression and trajectory of the frailty continuum.

OPTIMA-C will develop unifying administrative and data platforms, exploring the feasibility of inclusive screening for sarcopaenia early during rehabilitation hospital stay. Early muscle ultrasound will also be utilised to determine key muscles possibly predictive of rehabilitation functional or global outcomes in the studied populations and their correlation with acute disease outcomes. Digital markers are quantified and correlations are investigated with physical, muscle and bone imaging findings.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 50y
2. Asian ethnicity
3. First diagnosis (stroke, Traumatic Brain Injury (TBI), knee osteoarthritis, breast cancer)
4. Living in community
5. Able to understand 1 step simple commands
6. For inpatients: (i) within 12 weeks of disease (stroke/TBI) onset, and (ii) within 2 weeks of rehabilitation ward admission
7. For outpatients: (i) >6 months from initial diagnosis of first stroke, TBI, knee osteoarthritis or breast cancer, and (ii) at least standby assistance, modified independent or independent in ambulation with /without walking.

Exclusion Criteria:

1. Nursing home or dormitory resident
2. Non-resident status in Singapore (e.g. foreign worker, tourist, temporary visit pass)
3. Impairments affecting understanding of questionnaires and tasks: e.g. severe deafness, severe visual impairment and severe /global aphasia,
4. Presence of active fractures, dislocations, non-weight bearing status, burns, unhealed wounds, active skin infections/eczema and agitated behaviour or delirium
5. Anticipated life expectancy < 1 year
6. Presence of tracheostomy, ventilator, renal dialysis, end-organ failure
7. Patients with disorders of consciousness.
8. Pregnant or lactating participants

   For Knee Osteoarthritis patients only:
9. Alternative diagnosis to knee OA e.g. Referred pain from hip or spine.
10. Other forms of knee arthritis eg. Inflammatory, post traumatic
11. Previous knee arthroplasty

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in both outpatient and inpatient clinics
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Incidence (rates) of Frailty | Through study's data collection period, up to 4 years
  Based off different outcomes determined in the study
Severity of Frailty | For inpatient: Visit 1 (within 2 weeks of admission) to Visit 6 (end of 3rd year); For outpatient: Visit 1 (baseline) to Visit 4 (end of 3rd year)
  Based on CFS - 9-point clinical assessment tool evaluating an individual's frailty status; maximum score: 9; higher score indicates increased frailty.

SECONDARY OUTCOMES:
Body Composition Analysis (BCA) | For inpatient: Visit 3 (6 months post-event) to Visit 6 (end of 3rd year); For outpatient: Visit 1 (baseline) to Visit 4 (end of 3rd year)
  Measured using weak electrical current passed from feet to estimate proportion of muscle, fat and water mass.
Short Physical Performance Battery (SPPB) | For inpatient: Visit 1 (within 2 weeks of admission) to Visit 6 (end of 3rd year); For outpatient: Visit 1 (baseline) to Visit 4 (end of 3rd year)
  Measures 3 components: (1) 5 times chair stand test; (2) Balance test; (3) Gait speed (4m walk test). Score from 0-12 with higher score indicating greater functional capacity.
Hand Grip Strength (kg) | For inpatient: Visit 1 (within 2 weeks of admission) to Visit 6 (end of 3rd year); For outpatient: Visit 1 (baseline) to Visit 4 (end of 3rd year)
  Measured seated with arms on a table bent to 90° using a dynamometer (mean of 3 readings will be recorded)
Muscle Ultrasound imaging | For Inpatient: Visit 1 (within 2 weeks of admission), Visit 2 (1 week pre-discharge)
  Determines state of muscle health of arm, thigh and jaw muscles through size, area and structural properties.
FRAIL Questionnaire | For inpatient: Visit 1 (within 2 weeks of admission) to Visit 6 (end of 3rd year); For outpatient: Visit 1 (baseline) to Visit 4 (end of 3rd year)
  5-point questionnaire; (1-2 point) indicates pre-frail, (3-5 points) indicates frail

CONTACTS AND LOCATIONS:
Overall Officials: Karen Chua, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tay MRJ, Kim JM, Ong PL, Khin LW, Wong CJ, Kong KH, Tan BY, Lee ES, Sim SZ, Lim WS, Yam MGJ, Chew JL, Tan AWK, Sidarta A, Yee E, Chua KSG. Targeting osteosarcopenia and multimorbidity for frailty prevention through identification and deep phenotyping methods in healthy ageing and high-burden disease cohorts (OPTIMA-C): a longitudinal observational cohort study protocol for neuromusculoskeletal muscle health. BMJ Open. 2025 May 23;15(5):e094279. doi: 10.1136/bmjopen-2024-094279. PMID 40409965